CLINICAL TRIAL: NCT06561412
Title: A Pilot Randomized Trial of a Produce Prescription Intervention to Improve Health Among Food Insecure Adults With Chronic Kidney Disease
Brief Title: Penn Produce Prescription and Chronic Kidney Disease Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 855783
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Renal Insufficiency, Chronic; Food Insecurity
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: At the end of the baseline assessment, participants will be randomized using a permuted block technique with block size of 4 to either usual care (Arm 1) or to the produce prescription intervention (Arm 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will not receive the produce prescription vouchers but will still receive compensation for completing different study related tasks and will receive their usual medical care.
- Produce Prescription (Experimental): Participants will receive either $40 (families of 2 members or less) or $60 (families of more than 2 members) produce vouchers every 2 weeks for 6 months, for a total of $480 or $720. They will also receive compensation for completing different study related tasks and will receive their usual medical care.
  Interventions: Behavioral: Produce Prescription

INTERVENTIONS:
Behavioral: Produce Prescription — Participants will receive either $40 (families of 2 members or less) or $60 (families of more than 2 members) produce vouchers every 2 weeks for 6 months, for a total of $480 or $720. These vouchers are sponsored by The Food Trust.
  Arms: Produce Prescription

SUMMARY:
The goal of this pilot clinical trial is to examine the feasibility, acceptability, and likely effect of a produce prescription intervention on patient-centered outcomes, health behaviors and health outcomes, among food insecure adults with chronic kidney disease stages 3 - 5.

Participants will complete surveys at three timepoints, each three months apart, and complete health measurements at two timepoints 6 months apart. Half of the participants will be randomly assigned to the treatment where they will receive produce prescriptions with amount of the vouchers depending on their reported family size, every two weeks over six months. Researchers will compare the treatment group and the control group to see if there are any improvements in patient-centered outcomes (food and nutrition insecurity, health-related quality of life, depression and anxiety) and clinical outcomes (diet quality, metabolic acidosis, serum albumin, estimated GFR, blood pressure, and HbA1C).

DETAILED DESCRIPTION:
The study team will conduct a two-arm 1:1 randomized controlled trial to examine the feasibility, acceptability, and likely effect of a produce prescription intervention on patient-centered outcomes, health behaviors and health outcomes, among food insecure adults with CKD stages 3-5. The study's specific aims are:

Aim 1: Establish a community advisory board (CAB) to inform and guide the produce prescription intervention. The CAB will include patients, community members, CKD providers and relevant community partners.

Aim 2: Evaluate the effectiveness of a produce prescription intervention on clinical and patient centered outcomes in a randomized trial among (n=100) people with CKD and food insecurity. People with CKD stages 3-5 and food insecurity will be randomized to either a control or intervention group, which will receive a twice monthly produce prescription voucher to purchase fruits and vegetables at local stores for 6 months. Participants will be followed for patient-centered outcomes (food and nutrition insecurity, health-related quality of life, depression, and anxiety) and clinical outcomes (diet quality, metabolic acidosis, serum albumin, estimated GFR, blood pressure, and HbA1c). The study's hypothesis is that participants receiving the intervention will have improvements in food and nutrition security, diet quality and other patient-centered outcomes compared to the control group. The CKD clinical outcomes are exploratory and will serve as a proof-of-concept for this type of intervention in a CKD population.

Aim 3: Determine intervention acceptability and uptake and explore patient experiences with managing food insecurity and CKD. Researchers will administer surveys to eligible individuals who decline study enrollment (n=20), monitor self-report of voucher delivery and usage, and track voucher redemption rates to assess acceptability and uptake. Researchers will also conduct in-depth semi-structured interviews with participants in the intervention (n=20) and control (n=10) group to elucidate the experience of food insecurity and CKD co-management, coping strategies, and perceptions of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Lives within 5 miles of Philadelphia
* At least one recent clinic visit at Penn Renal Care, or one clinic visit at Penn Primary Care (earliest six months before start of recruitment)
* Positive screening of food insecurity in the electronic health record (EHR) within the prior 2 months
* Diagnosis of chronic kidney disease stages 3 -5

Exclusion Criteria:

* Does not meet all of the inclusion criteria
* Unable to provide consent
* Non-English speaker
* Cognitive impairment, per principal investigators' discretion
* Marked as "do not contact" in EMR for research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in food insecurity category | Assessed via survey at baseline, 3 months, and 6 months.
  Change from baseline in food insecurity in the last 30 days as measured by USDA Household Food Security six-item short form survey. Outcome is 3 ordered categories: high or marginal food insecurity (score 0-1 on the scale), low food security (score 2 -4 on the scale), very low food security (score 5 -6 on the scale). The minimum score is 0, and the maximum score is 6.
Change in nutritional security sore | Assessed via survey at baseline, 3 months, and 6 months.
  Change from baseline in nutrition security score in the last 30 days as measured by the Center for Nutrition & Health Impact Nutrition Security Scale. Outcome is continuous (scores 0-4). Higher scores indicate a higher degree of household nutritional security.
Change in fruit and vegetable consumption | Assessed via survey at baseline, 3 months, and 6 months.
  Change from baseline in fruit and vegetable consumption in the last month as measured by a food frequency questionnaire. Outcomes are ordered by frequency/quantity over the time period.

SECONDARY OUTCOMES:
Change in anxiety category | Assessed via survey at baseline, 3 months, and 6 months.
  Change from baseline in anxiety category in the last two weeks as measured by the Primary Care Evaluation of Mental Health Disorders Patient Health Questionnaire's GAD-7 Anxiety survey. Outcome is ordered in 4 categories: minimal anxiety (score 0-4 on the scale), mild anxiety (score 5-9 on the scale), moderate anxiety (score 10-14 on the scale), severe anxiety (score 15-21 on the scale).
Change in depression category | Assessed via survey at baseline, 3 months, and 6 months.
  Change from baseline in depression category in the last two weeks as measured by the Patient Health Questionnaire (PHQ-9). Outcome is ordered in 5 categories: none to minimal depression (score 0-4 on the scale), mild depression (score 5-9 on the scale), moderate depression (score 10-14 on the scale), moderately severe depression (score 15-18 on the scale), severe depression (score 20-27 on the scale).
Change in kidney disease quality of life | Assessed via survey at baseline, 3 months, and 6 months.
  Change from baseline in kidney disease quality of life in the last four weeks as measured by the Kidney Disease and Quality of Life (KDQOL-36) survey. Outcome is ordered in 3 categories: above average, average, and below average, compared to others of the same age, gender, and diabetes status. The scale scores the patient from 0-100, with higher scores indicating higher health-related quality of life.
Serum albumin | Assessed via blood draw at baseline and 6 months
  Change from baseline in serum albumin
Metabolic acidosis | Assessed via blood draw at baseline and 6 months
  Change from baseline in bicarbonate level
Estimated Glomerular Filtration Rate (eGFR) | Assessed at baseline and 6 months
  Change from baseline in eGFR
Blood Pressure | Assessed at baseline and 6 months
  Change from baseline in blood pressure
Hemoglobin A1c | Assessed at baseline and 6 months
  Change from baseline in HBA1c; only measured in participants diagnosed with diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Kinsey, PhD, MPH, Principal Investigator — University of Pennsylvania; Sarah Schrauben, MD, MSCE, Principal Investigator — University of Pennsylvania; Nandta Mitra, PhD, Principal Investigator — University of Pennsylvania; Stefanie Hinkle, PhD, Principal Investigator — Assistant Professor of Epidemiology, Departments of Biostatistics, Epidemiology and Informatics
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No